CLINICAL TRIAL: NCT01758497
Title: Fascia Iliaca Compartment Block For Analgesia After Total Hip Arthroplasty; A Randomized Double Blind, Placebo-Controlled Trial
Brief Title: Fascia Iliaca Compartment Block For Analgesia After Total Hip Arthroplasty
Acronym: FICB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-042
Record Dates: First submitted 2012-06-06; First posted 2013-01-01 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Pain Disorder; Sensory Deficit
Keywords: Fascia Iliaca compartment block, Pain, Sensorial blockade
MeSH Terms: conditions — Somatoform Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Active Comparator): US guided injections of 30 ml 0.5% ropivacaine (Fascia Iliaca Compartment Block)
  Interventions: Procedure: Fascia iliaca compartment block
- Saline (Sham Comparator): US guided injections of 30 ml 0.9% NaCl (Fascia Iliaca Compartment Block)
  Interventions: Procedure: Fascia Iliaca compartment block

INTERVENTIONS:
Procedure: Fascia iliaca compartment block — 30 ml 0.5% ropivacaine, beneath the fascia iliaca
  Other Names: Ultrasound guided Fascia iliaca compartment block; FICB
  Arms: Ropivacaine
Procedure: Fascia Iliaca compartment block — 30 ml 0.9% NaCl (sham block, SB), beneath the fascia iliaca
  Other Names: Ultrasound guided Fascia iliaca compartment block; FICB
  Arms: Saline

SUMMARY:
Introduction Fascia Iliaca compartment block (FICB) is commonly used to treat pain in patients after total hip arthroplasty (THA) despite the lack of RCTs to evaluate the efficacy of FICB for this indication. Therefore the objective of this study was to assess the analgesic benefit of FICB for post-operative pain management in THA.

Methods After IRB approval and informed consent, patients having THA at our center in the period 2010-2011 were recruited. Eligible patients were adults, ASA physical status I-III, and BMI <30) with no contraindication to study procedures. In the PACU, all patients received morphine sulfate IVPCA; patients reporting pain > 3 on the NRS-11 despite IVPCA were randomized by the method of sealed envelopes to receive US guided injections of 30ml 0.5% ropivacaine (FICB) or 30ml 0.9% NaCl (sham block, SB) beneath the fascia iliaca.

The primary outcome variable was opioid analgesic consumption during the first 24 h postoperatively. Secondary outcome measures were pain intensity (NRS-11) and extent of sensory blockade.

DETAILED DESCRIPTION:
Introduction Fascia Iliaca compartment block (FICB) is commonly used to treat pain in patients after total hip arthroplasty (THA) despite the lack of RCTs to evaluate the efficacy of FICB for this indication. Therefore the objective of this randomized, prospective trial was to assess the analgesic benefit of FICB for post-operative pain management in THA. Our hypothesis was that FICB would confer an analgesic benefit for patients after THA.

Methods After IRB approval and informed consent, patients having THA at our center in the period 2010-2011 were recruited in the morning of their surgery. Eligible patients were adults, ASA physical status I-III, and BMI <30) with no contraindication to study procedures. In the PACU, all patients received morphine sulfate IVPCA; patients reporting pain > 3 on the NRS-11 despite IVPCA were randomized by the method of sealed envelopes to receive US guided injections of 30ml 0.5% ropivacaine (FICB) or 30ml 0.9% NaCl (sham block, SB) beneath the fascia iliaca.

The primary outcome variable was opioid analgesic consumption during the first 24 h postoperatively. Secondary outcome measures were pain intensity (NRS-11) and extent of sensory blockade.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* ASA physical status I-III
* BMI<30
* No contraindications to study procedures

Exclusion Criteria:

* Pediatric patients
* ASA physical status IV
* BMI>30
* Contraindications to study procedures
* Hypersensitivity to local anesthetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic consumption | 24 h postoperatively

SECONDARY OUTCOMES:
Pain intensity (NRS-11) and extent of sensory blockade | 24 h postoperatively
  Pain intensity was assessed immediately before and after block placement and at 10-min intervals for the first 30 min after block. Sensory assessment was at 30 min after block, using a pinprick test in the lateral, medial and anterior aspects of the thigh. Specifically, sensation in the territories of the lateral femoral cutaneous, obturator, and femoral nerves was tested using a scale of 0-2 ( 0 = no sensation, 1 = diminished sensation, 2= full sensation). Assessment of motor blockade was not possible because of lower extremity immobilization after surgery to prevent hip dislocation.

CONTACTS AND LOCATIONS:
Overall Officials: Admir Hadzic, MD,PhD, Study Director — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St Luke's Roosevelt Hospitals, New York, New York, United States

REFERENCES:
- [Result] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Result] Dolan J, Williams A, Murney E, Smith M, Kenny GN. Ultrasound guided fascia iliaca block: a comparison with the loss of resistance technique. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):526-31. doi: 10.1016/j.rapm.2008.03.008. PMID 19258967
- [Result] Weller RS. Does fascia iliaca block result in obturator block? Reg Anesth Pain Med. 2009 Sep-Oct;34(5):524; author reply 524. doi: 10.1097/AAP.0b013e3181ada59f. No abstract available. PMID 19749590
- [Result] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Result] Stevens M, Harrison G, McGrail M. A modified fascia iliaca compartment block has significant morphine-sparing effect after total hip arthroplasty. Anaesth Intensive Care. 2007 Dec;35(6):949-52. doi: 10.1177/0310057X0703500615. PMID 18084988
- [Result] Goitia Arrola L, Telletxea S, Martinez Bourio R, Arizaga Maguregui A, Aguirre Larracoechea U. [Fascia iliaca compartment block for analgesia following total hip replacement surgery]. Rev Esp Anestesiol Reanim. 2009 Jun-Jul;56(6):343-8. doi: 10.1016/s0034-9356(09)70406-2. Spanish. PMID 19725341
- [Result] Biboulet P, Morau D, Aubas P, Bringuier-Branchereau S, Capdevila X. Postoperative analgesia after total-hip arthroplasty: Comparison of intravenous patient-controlled analgesia with morphine and single injection of femoral nerve or psoas compartment block. a prospective, randomized, double-blind study. Reg Anesth Pain Med. 2004 Mar-Apr;29(2):102-9. doi: 10.1016/j.rapm.2003.11.006. PMID 15029544